CLINICAL TRIAL: NCT07323927
Title: An Investigator Initiated Trial Evaluating the Therapeutic Efficacy of Galcanezumab in Patients With Alzheimer's Disease
Brief Title: Investigator Initiated Trial of Galcanezumab Treatment in Alzheimer's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025162
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Galcanezumab
MeSH Terms: conditions — Alzheimer Disease | interventions — galcanezumab; erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Galcanezumab Treatment Arm (Open-label) (Experimental): Subcutaneous Galcanezumab administration with an initial dose of 240 mg (single injection), followed by 120 mg every 4 weeks for a total of 6 doses (24-week treatment duration).
  Interventions: Drug: Galcanezumab

INTERVENTIONS:
Drug: Galcanezumab — Subcutaneous injection; monotherapy (administered at the designated study site: Advanced Innovation Center for Neurological Disorders, Xuanwu Hospital, Capital Medical University); initial dose: 240 mg (single administration) followed by 120 mg every 4 weeks for 6 total doses
  Other Names: Emgality

SUMMARY:
This single-arm, open-label clinical study systematically evaluates the efficacy and safety of Galcanezumab in patients with mild-to-moderate Alzheimer's disease (AD). Eligible participants who provided written informed consent were screened and enrolled to receive Galcanezumab treatment. The therapeutic regimen involved subcutaneous administration of Galcanezumab with an initial 240 mg loading dose followed by 120 mg maintenance doses every four weeks for six total administrations over a 24-week treatment period. All study procedures were conducted at the Advanced Innovation Center for Neurological Disorders, Xuanwu Hospital, Capital Medical University. Comprehensive data collection and clinical assessments were performed at baseline (pre-treatment), week 12 (Visit 3), week 24 (Visit 4), and week 36 (Visit 5, 12 weeks after the final dose) to evaluate treatment outcomes and safety profiles. The study design incorporates standardized clinical trial methodology while maintaining the flexibility required for exploratory therapeutic evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50 and 90 years at enrollment, regardless of gender;
2. Meeting the NIA-AA core clinical criteria for probable Alzheimer's disease;
3. Clinical Dementia Rating - Global Score (CDR-GS) between ≥1 and ≤2; Clinical Dementia Rating - Memory Box (CDR-Memory box) ≥0.5;
4. Amyloid PET or cerebrospinal fluid (CSF) biomarkers consistent with AD pathology;
5. Mini-Mental State Examination (MMSE) score between ≥12 and ≤26;
6. Non-illiterate or with at least 4 to 6 years of formal education;
7. If currently taking psychiatric or cognitive-enhancing medications, the dosage must have been stable for at least 3 months prior to the study and remain unchanged during the study. Unless otherwise specified, all permitted concomitant medications (non-AD related) must have been stable for at least 4 weeks prior to baseline;
8. Availability of a reliable caregiver or legal guardian able to support the participant throughout the study, defined as spending at least 8 hours per week with the participant;
9. Willingness to participate in the clinical trial, maintain existing interventions during the study period, and provision of signed informed consent.

Exclusion Criteria:

1. Presence of neuropsychiatric symptoms outside the typical spectrum of Alzheimer's disease;
2. History of transient ischemic attack (TIA), stroke, or seizure within the past 12 months;
3. Known allergy to gantenerumab or its excipients, or severe allergic reactions to monoclonal antibodies;
4. Cardiovascular or gastrointestinal diseases including severe arrhythmias, uncontrolled hypertension (systolic >180 mmHg or diastolic >110 mmHg), or active peptic ulcer disease, inflammatory bowel disease, or other conditions likely to exacerbate gastrointestinal adverse reactions;
5. MRI contraindications such as cardiac pacemaker/defibrillator or ferromagnetic metal implants;
6. MRI evidence of other clinically significant lesions suggesting dementia diagnoses other than AD;
7. MRI findings of other important pathologies, including but not limited to: single hemorrhagic lesions >10 mm in diameter; evidence of vasogenic edema; brain contusions, softening, aneurysms, vascular malformations, or infectious lesions; strokes involving major vascular territories; severe small vessel or white matter disease; space-occupying lesions; or brain tumors (meningiomas or arachnoid cysts with a maximum diameter <1 cm may be allowed);
8. Current participation in another clinical trial targeting AD improvement;
9. Any unstable or inadequately controlled medical condition, or other situations deemed by investigators to compromise participant safety or study assessments;
10. Other investigator-determined reasons precluding participant inclusion.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
CGRP Levels in Cerebrospinal Fluid and Plasma | Baseline; 24 weeks.
  Measurement of CGRP levels in cerebrospinal fluid and plasma.

SECONDARY OUTCOMES:
Change from baseline on the Alzheimer's disease assessment scale-cognitive section(ADAS-Cog) | baseline; 12 weeks; 36 weeks.
Change from baseline on the Alzheimer's disease assessment scale-cognitive section(ADAS-Cog) | baseline; 24 weeks.
Change from baseline on the Mini Mental state Examination (MMSE) score | baseline; 12 weeks; 24 weeks; 36 weeks.
Change from baseline on the Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) | baseline; 12 weeks; 24 weeks; 36 weeks.
Change from baseline on the Alzheimer's Disease Cooperative study-clinical global impression of change scale(ADCS-CGIC) | baseline; 12 weeks; 24 weeks; 36 weeks.
Change from baseline on the Alzheimer's Disease Cooperative study-Activities of Daily Living Scale(ADCS-ADL) | baseline; 12 weeks; 24 weeks; 36 weeks.
Change from baseline on the Neuropaychiatic Inventory (NPI) | baseline; 12 weeks; 24 weeks; 36 weeks
Change from baseline on the Hamilton depression scale (HAMD) | baseline; 12 weeks; 24 weeks; 36 weeks
Change from baseline in amplitude of Low-Frequency Fluctuations (ALFF) in resting-state functional MRI | baseline; 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, Study Chair — M.D., Ph.D.
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No